CLINICAL TRIAL: NCT06245317
Title: Effects of Pressure Controlled-volume Guarantee Ventilation on Respiratory Mechanics in Pediatric Laparoscopic Surgery
Brief Title: PCV-VG in Pediatric Laparoscopic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Muhammed Mahmoud Khalil, Resident Physician, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 04-2023-200588
Record Dates: First submitted 2024-01-14; First posted 2024-02-07 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia Complication; Mechanical Ventilation Complication

STUDY DESIGN:
Intervention Model Description: effects of Pressure Controlled Ventilation - Volume Guarantee (PCV-VG) mode with volume control ventilation (VCV) and pressure control ventilation (PCV) modes on respiratory mechanics (including the dynamic compliance, PIP, mean airway pressure, driving pressure..etc) and oxygenation in paediatrics laparoscopic surgery.
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pressure control ventilation-volume guarantee (PCV-VG) group (Active Comparator): In the PCV-VG group the tidal volume will be set to 8-10ml/kg and the respiratory rate will be adjusted according to oxygen saturation and end-tidal CO¬2.
  Interventions: Device: Mechanical Ventilation Mode
- Pressure control ventilation (PCV) group (Active Comparator): In the PCV group peak inspiratory pressure will be set to 10-15 cm H2O titrated to achieve 8-10 ml/kg and the respiratory rate will be adjusted according to oxygen saturation and end-tidal Co2
  Interventions: Device: Mechanical Ventilation Mode
- Volume control ventilation (VCV) group (Active Comparator): In the VCV group tidal volume will be set to 8-10 ml/kg and the respiratory rate will be adjusted according to oxygen saturation and end-tidal CO2,
  Interventions: Device: Mechanical Ventilation Mode

INTERVENTIONS:
Device: Mechanical Ventilation Mode — Each arm will have a different ventilation mode according to the allocation.

SUMMARY:
This Study will aim to compare the effects of Pressure Controlled Ventilation - Volume Guarantee (PCV-VG) mode with volume control ventilation (VCV) and pressure control ventilation (PCV) modes on respiratory mechanics (including the dynamic compliance, PIP, mean airway pressure, driving pressure..etc) and oxygenation in pediatric laparoscopic surgery.

DETAILED DESCRIPTION:
Laparoscopic surgery is superior to open surgery in terms of recovery time, less postoperative pain, less wound complications, shorter hospital stay, and earlier return to work. However, carbon dioxide insufflation causes several intraoperative cardiovascular, renal, and respiratory adverse effects. Regarding respiratory effects, elevated Intra-abdominal pressure and abdominal expansion shifts the diaphragm upwards. Thus, intrathoracic pressure increases, and expansion of the lungs is restricted. This is followed by a significant decrease up to 50% in pulmonary dynamic compliance and an increase in peak and plateau airway pressures. After deflation of pneumoperitoneum both the pulmonary compliance and airway pressures return to the baseline levels. High airway pressures and decreased compliance can be associated with pulmonary barotrauma, which may manifest as immediate pneumothorax. The basal lung regions are compressed during elevated IAP causing atelectasis and uneven ventilation-perfusion relationships, impairing gas exchange. Hence, the choice of ventilation mode is very important, especially in the paediatric population. Volume control ventilation (VCV) and pressure control ventilation (PCV) modes have been used but each has its own drawbacks, with the former risking increase in airway pressure when pulmonary compliance changes which can lead to barotrauma and the latter not guaranteeing the desired tidal volume which leads to hypoventilation that presents with hypercarbia. Pressure Control Ventilation - Volume Guarantee (PCV-VG) is a recent controlled ventilation mode that combines the benefits of both volume control ventilation (VCV) and pressure control ventilation (PCV) by delivering the preset tidal volume with a decelerating flow at the lowest possible peak inspiratory pressure during a preset inspiratory time and at a preset respiratory rate ensuring adequate ventilation .

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II.
* Both sexes.
* Age: 1-8 years old.
* Scheduled for elective abdominal or urologic laparoscopic surgery.
* BMI between the 5th and 95th percentiles.

Exclusion Criteria:

* ASA physical status more than II.
* Pre-existing lung disease.
* Pre-operative chest infection.
* Any thoracic deformities.
* Unsatisfactory pre-operative arterial oxygen saturation or haemoglobin level.
* Patients with cardiac, hepatic, or renal diseases.
* BMI above and below the 95th and 5th percentile respectively.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Lung dynamic compliance (Cdyn) | 5 minutes after intubation (T1), 5 minutes after pneumoperitoneum (T2), 15 minutes after pneumoperitoneum (T3), 5 minutes after desufflation of pneumoperitoneum (T4) and 5 minutes after the operation (T5)
  Dynamic compliance represents pulmonary compliance during periods of gas flow, such as during active inspiration.

SECONDARY OUTCOMES:
PaO2 | 5 minutes after intubation (T1), 5 minutes after pneumoperitoneum (T2), 15 minutes after pneumoperitoneum (T3), 5 minutes after desufflation of pneumoperitoneum (T4) and 5 minutes after the operation (T5)
  The PaO2 partial pressure from arterial blood gas analysis will be recorded.
SpO2% | 5 minutes after intubation (T1), 5 minutes after pneumoperitoneum (T2), 15 minutes after pneumoperitoneum (T3), 5 minutes after desufflation of pneumoperitoneum (T4) and 5 minutes after the operation (T5)
  The peripheral arterial saturation will be recorded.
PaCO2 | 5 minutes after intubation (T1), 5 minutes after pneumoperitoneum (T2), 15 minutes after pneumoperitoneum (T3), 5 minutes after desufflation of pneumoperitoneum (T4) and 5 minutes after the operation (T5)
  The PaCo2 partial pressure from arterial blood gas analysis will be recorded.
End-tidal CO2 | 5 minutes after intubation (T1), 5 minutes after pneumoperitoneum (T2), 15 minutes after pneumoperitoneum (T3), 5 minutes after desufflation of pneumoperitoneum (T4) and 5 minutes after the operation (T5)
  The end-tidal CO2 will be recoded from the main stream capnography
Mean airway pressure | 5 minutes after intubation (T1), 5 minutes after pneumoperitoneum (T2), 15 minutes after pneumoperitoneum (T3), 5 minutes after desufflation of pneumoperitoneum (T4) and 5 minutes after the operation (T5)
  The mean airway pressure will be recorded from the ventilator electronic display in the GE anesthesia machine
Peak inspiratory pressure | 5 minutes after intubation (T1), 5 minutes after pneumoperitoneum (T2), 15 minutes after pneumoperitoneum (T3), 5 minutes after desufflation of pneumoperitoneum (T4) and 5 minutes after the operation (T5)
  The PIP will be recorded from the ventilator electronic display in the GE anesthesia machine
Tidal volume | 5 minutes after intubation (T1), 5 minutes after pneumoperitoneum (T2), 15 minutes after pneumoperitoneum (T3), 5 minutes after desufflation of pneumoperitoneum (T4) and 5 minutes after the operation (T5)
  The exhaled tidal volume will be recorded from the ventilator electronic display in the GE anesthesia machine

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Study Director — Assiut University; Yara H Abbas, MD, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No